CLINICAL TRIAL: NCT04834843
Title: Temporal Trends in the Incidence, Treatment Patterns, and Outcomes of COronary Artery Disease and PEripheral Artery Disease (COPE) in Korea
Brief Title: Temporal Trends of COronary Artery Disease and PEripheral Artery Disease (COPE) in Korea
Acronym: COPE registry
Status: Completed | Type: Observational
Sponsor: Wonju Severance Christian Hospital (Other)
Responsible Party: Principal Investigator, Dong-Hyuk Cho, Assistant professor, Wonju Severance Christian Hospital
Other Study IDs: 2020AN0279
Record Dates: First submitted 2021-04-05; First posted 2021-04-08 (Actual); Last update posted 2021-04-08 (Actual); Status verified 2021-04

CONDITIONS: Coronary Artery Disease; Peripheral Artery Disease; Cardiovascular Diseases
MeSH Terms: conditions — Coronary Artery Disease; Peripheral Arterial Disease; Cardiovascular Diseases | interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Observational study, no intervention — Observational study, no intervention

SUMMARY:
Cardiovascular disease (CVD) is caused by atherosclerosis of the artery and is classified into coronary artery disease, cerebrovascular disease, and peripheral arterial disease, depending on the location of the artery and the target organs. However, since CVD share a similar pathophysiology and the probability of incidence of other CVD in CVD patients is very high. It is thought that CVD incidence and mortality can be reduced by predicting the degree of incidence of other CVD in CVD patients. The aim of this study is to investigate the incidence and mortality of other CVD diseases in CVD patients.

ELIGIBILITY:
Inclusion Criteria:

* Koreans who diagnosed with coronary artery disease between 2009 and 2018
* Koreans who diagnosed with peripheral artery disease between 2009 and 2018
* Koreans who diagnosed with cerebrovascular disease between 2009 and 2018
* more than 18 years old

Exclusion Criteria:

* less than 18 years old

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: People aged at least 18 years old with CAD, PAD, or cerebrovascular disease were identified from Korean national health insurance using International Classification of Diseases, tenth revision (ICD-10) codes.
Sampling Method: Probability Sample
Enrollment: 700000 (Actual)
Dates: Start 2009-01-01 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Incidence of coronary artery disease, cerebrovascular disease, peripheral arterial disease | Up to 10 years
  Among all Koreans, percentage (%) of patients with a history of being diagnosed with CVD and underwent in-hospital treatment

SECONDARY OUTCOMES:
1-year mortality | Up to 1 year
  The percentage (%) of any CVD related mortality

IPD SHARING:
Plan to Share IPD: No
The IPD from Korean national health insurance is not publicly accessible due to Korean personal information projection act

REFERENCES:
- [Result] Sundaram V, Bloom C, Zakeri R, Halcox J, Cohen A, Bowrin K, Briere JB, Banerjee A, Simon DI, Cleland JGF, Rajagopalan S, Quint JK. Temporal trends in the incidence, treatment patterns, and outcomes of coronary artery disease and peripheral artery disease in the UK, 2006-2015. Eur Heart J. 2020 May 1;41(17):1636-1649. doi: 10.1093/eurheartj/ehz880. PMID 31883328
- [Result] Bhatt DL, Steg PG, Ohman EM, Hirsch AT, Ikeda Y, Mas JL, Goto S, Liau CS, Richard AJ, Rother J, Wilson PW; REACH Registry Investigators. International prevalence, recognition, and treatment of cardiovascular risk factors in outpatients with atherothrombosis. JAMA. 2006 Jan 11;295(2):180-9. doi: 10.1001/jama.295.2.180. PMID 16403930
- [Result] Ahn S, Park YJ, Min SI, Kim SY, Ha J, Kim SJ, Kim HS, Yoon BW, Min SK. High prevalence of peripheral arterial disease in Korean patients with coronary or cerebrovascular disease. J Korean Med Sci. 2012 Jun;27(6):625-9. doi: 10.3346/jkms.2012.27.6.625. Epub 2012 May 26. PMID 22690093
- [Result] Sogaard M, Nielsen PB, Skjoth F, Eldrup N, Larsen TB. Temporal Changes in Secondary Prevention and Cardiovascular Outcomes After Revascularization for Peripheral Arterial Disease in Denmark: A Nationwide Cohort Study. Circulation. 2021 Mar 2;143(9):907-920. doi: 10.1161/CIRCULATIONAHA.120.047994. Epub 2020 Dec 10. PMID 33300375